CLINICAL TRIAL: NCT03792217
Title: Postoperative Pain After Endodontic Irrigation Using 1.3% Versus 5.25% Sodium Hypochlorite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Suzan AW Amin, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ENDO-CU-2011-7-25
Record Dates: First submitted 2018-12-24; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Dental Pulp Necrosis
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.3% NaOCl (Experimental): Root canal irrigation done using 1.3% NaOCl.
  Interventions: Other: 1.3% NaOCl
- 5.25% NaOCl (Active Comparator): Root canal irrigation done using 5.25% NaOCl.
  Interventions: Other: 5.25% NaOCl

INTERVENTIONS:
Other: 1.3% NaOCl — Endodontic irrigant
  Other Names: 1.3% sodium hypochlorite
  Arms: 1.3% NaOCl
Other: 5.25% NaOCl — Endodontic irrigant
  Other Names: 5.25% sodium hypochlorite
  Arms: 5.25% NaOCl

SUMMARY:
The aim of this prospective, randomized, clinical trial was to evaluate the effect of 1.3% sodium hypochlorite (NaOCl) concentration versus 5.25% NaOCl concentration on post-operative pain and medication intake in adult patients with pulp necrosis in mandibular molars.

DETAILED DESCRIPTION:
The aim of this prospective, randomized, clinical trial was to evaluate the effect of 1.3% sodium hypochlorite (NaOCl) concentration versus 5.25% NaOCl concentration on post-operative pain and medication intake in adult patients with pulp necrosis in mandibular molars. Medical and dental history was obtained from all participants in this trial and clinical and radiographic evaluation for teeth was recorded. Participants with pulp necrosis with or without apical periodontitis were included. After access cavity preparation, participants were randomly assigned to one of the following groups: experimental group (irrigation using 1.3% NaOCl) or control group (irrigation using 5.25% NaOCl ). Two-visit root canal treatment was performed with a week interval in between visits. Each patient received a 7-day diary to record postoperative pain and rescue medication intake. Post-operative pain was measured at the following time points: immediately , 3, 24, 48 hours and 7 days after the first visit and postobturation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 25-45 year old.
2. Medically free.
3. Non-vital mandibular teeth (first or second molar) with or without apical periodontitis
4. No sex predilection

Exclusion Criteria:

1. Pregnant females.
2. History of allergy to any medication used in the study.
3. Preoperative premedication 12 hours before procedure.
4. Acute abscess cases.
5. Badly-decayed crown.
6. Retreatment cases

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 308 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain using a pain-measuring scale | immediately after treatment
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured immediately after the first visit
Postoperative pain using a pain-measuring scale | 3 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 3 hours after the first visit
Postoperative pain using a pain-measuring scale | 24 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 24 hours after the first visit
Postoperative pain using a pain-measuring scale | 48 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 48 hours after the first visit
Postoperative pain using a pain-measuring scale | 7 days
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 7 days after the first visit
Postoperative pain using a pain-measuring scale | immediately after obturation
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured immediately after obturation.

SECONDARY OUTCOMES:
Sham medication intake incidence | 7 days
  Sham medication intake incidence (Yes/No) taken as an initial rescue medication in case of postoperative pain.
Analgesic medication intake incidence | 7 days
  Analgesic medication intake incidence (Yes/No) as a rescue medication in case postoperative pain persisted after the sham medication intake.

CONTACTS AND LOCATIONS:
Overall Officials: Suzan Amin, PhD, Study Director — Cairo University; Randa El-Boghdady, PhD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Almeida G, Marques E, De Martin AS, da Silveira Bueno CE, Nowakowski A, Cunha RS. Influence of irrigating solution on postoperative pain following single-visit endodontic treatment: randomized clinical trial. J Can Dent Assoc. 2012;78:c84. PMID 22985896
- [Background] Bashetty K, Hegde J. Comparison of 2% chlorhexidine and 5.25% sodium hypochlorite irrigating solutions on postoperative pain: a randomized clinical trial. Indian J Dent Res. 2010 Oct-Dec;21(4):523-7. doi: 10.4103/0970-9290.74225. PMID 21187618
- [Background] Farzaneh S, Parirokh M, Nakhaee N, Abbott PV. Effect of two different concentrations of sodium hypochlorite on postoperative pain following single-visit root canal treatment: a triple-blind randomized clinical trial. Int Endod J. 2018 Jan;51 Suppl 1:e2-e11. doi: 10.1111/iej.12749. Epub 2017 Mar 6. PMID 28134983